CLINICAL TRIAL: NCT03578770
Title: Safety and Efficacy of the New 20 mm Lumen Apposing Metal Stent (Lams) for Endoscopic Treatment of Pancreatic and Peripancreatic Fluid Collections: a Large, International, Multicenter Study
Brief Title: Safety and Efficacy of the New 20 mm Lumen Apposing Metal Stent (Lams) for Endoscopic Treatment of Pancreatic and Peripancreatic Fluid Collections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: Axios 20 mm
Record Dates: First submitted 2018-05-21; First posted 2018-07-06 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Pancreatic Diseases
MeSH Terms: conditions — Pancreatic Diseases

STUDY DESIGN:
Intervention Model Description: Feasibility device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Hot Axios stent — Hot Axios stent

SUMMARY:
Pancreatic fluid collections (PFC) can occur as a complication of acute and chronic pancreatitis. PFC include pancreatic pseudocysts (PP) and walled-off necrosis (WON).

The majorities of WON are asymptomatic and will resolve spontaneously. Endoscopic ultrasound (EUS)-guided drainage has become the preferred treatment in the management of symptomatic PFC, with significant advantages compared with surgical and percutaneous drainage. Successful endoscopic management of the pancreatic fluid collections depends on the type of PFC. Studies have shown that endoscopic drainage of PP is greater than 90%, while success for WON is at best between 50-65%. Differences in treatment outcome are attributed to the viscosity and debris content of the PFC. Traditionally, the EUS-guided drainage has been performed with placement of multiple plastic stents or fully covered self-expanding metal stent.

Recently, lumen-apposing metal stents (LAMS) have been developed. LAMS have been utilized for the access and drainage of pancreatic fluid collections (PFCs). To date, a variety of LAMS sizes have been commercially available and widely used. Studies have shown high technical success (89-100%) and high clinical success rate (93-100%). The larger diameter of LAMS facilitates better drainage of PFC contents when compared to the small caliber of plastic stents and allows necrosectomy in repeated sessions without the need for stent replacement.

A new LAMS with a larger (20mm) lumen diameter (the Hot Axios, Boston Scientific, Natick MA, USA) was released on the market, with the idea that a larger diameter would allow a faster drainage of PFCs and facilitate endoscopic necrosectomy. This is currently the largest diameter LAMS available.

Further studies are needed to determine the ideal size for a LAMS going forward to achieve maximal clinical benefit with minimal patient risk.

Aim of the investigator's study is to evaluate the safety and efficacy of the new 20 mm Hot Axios stent placement for EUS-guided transmural drainage of pancreatic fluid collections.

DETAILED DESCRIPTION:
Pancreatic fluid collections (PFC) can occur as a complication of acute and chronic pancreatitis. PFC include pancreatic pseudocysts (PP) and walled-off necrosis (WON).

The majorities of WON are asymptomatic and will resolve spontaneously. Endoscopic ultrasound (EUS)-guided drainage has become the preferred treatment in the management of symptomatic PFC, with significant advantages compared with surgical and percutaneous drainage. Successful endoscopic management of the pancreatic fluid collections depends on the type of PFC. Studies have shown that endoscopic drainage of PP is greater than 90%, while success for WON is at best between 50-65%. Differences in treatment outcome are attributed to the viscosity and debris content of the PFC. Traditionally, the EUS-guided drainage has been performed with placement of multiple plastic stents or fully covered self-expanding metal stent.

Recently, lumen-apposing metal stents (LAMS) have been developed. LAMS have been utilized for the access and drainage of pancreatic fluid collections (PFCs). To date, a variety of LAMS sizes have been commercially available and widely used. Studies have shown high technical success (89-100%) and high clinical success rate (93-100%). The larger diameter of LAMS facilitates better drainage of PFC contents when compared to the small caliber of plastic stents and allows necrosectomy in repeated sessions without the need for stent replacement.

A new LAMS with a larger (20mm) lumen diameter (the Hot Axios, Boston Scientific, Natick MA, USA) was released on the market, with the idea that a larger diameter would allow a faster drainage of PFCs and facilitate endoscopic necrosectomy. This is currently the largest diameter LAMS available.

Further studies are needed to determine the ideal size for a LAMS going forward to achieve maximal clinical benefit with minimal patient risk.

Aim of the investigator's study is to evaluate the safety and efficacy of the new 20 mm Hot Axios stent placement for EUS-guided transmural drainage of pancreatic fluid collections.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients who underwent EUS-guided 20 mm Hot Axios stent placement for PFCs were included.

Exclusion Criteria:

* No exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
The investigators will evaluate the use of the new 20 mm Hot Axios in endoscopic transmural drainage through the reduction pof the bilirubin's value | 24 months

SECONDARY OUTCOMES:
The investigators will assess the rate/severity of adverse events (AEs) (ASGE lexicon). | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Repici Alessandro, MD, Principal Investigator — Humanitas Research Hospital IRCCS, Rozzano-Milan
Locations (1):
- Humanitas Research Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: No